CLINICAL TRIAL: NCT06908473
Title: A Multicenter, Double-Blind, Randomized Controlled Study on the Impact of Tongmai Jiangtang Capsules on the Risk of Cardiovascular and Cerebrovascular Events in Metabolic Syndrome
Brief Title: Tongmai Jiangtang Capsule for Cardiovascular Clinical Outcomes in High-Risk Metabolic Syndrome Patients
Acronym: TORCH-met
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: TCM hospital of Sichuan Province (Unknown); Xiyuan Hospital of CACMS (Unknown); Shanxi Provincial hospital of Chinese Medicine (Unknown); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Yinchuan Brain-Heart Simultaneous Treatment Internet Hospital Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Zhenjie Liu, Doctor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZLiu
Record Dates: First submitted 2025-03-15; First posted 2025-04-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome; Cardiovascular Disease (CKD); Cerebrovascular Disease; Qi Deficiency and Blood Stasis
Keywords: Metabolic Syndrome; High Cardiovascular and Cerebrovascular Risk Metabolic Syndrome, HCR-MS; Qi-Deficiency and Blood Stasis Syndrome; Tongmai Jiangtang Capsule
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Cerebrovascular Disorders | interventions — Color; Dosage Forms; Weights and Measures; Taste

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Tongmai Jiangtang Capsule Group) (Experimental): Participants in this Arm will receive Tongmai Jiangtang Capsule (TJC) in addition to standard treatment.
  Dosage: Three capsules, three times daily (tid), taken orally. Duration: The intervention period is 26 weeks, followed by a 26-week follow-up. Objective: This Arm aims to evaluate the efficacy of TJC in reducing cardiovascular and cerebrovascular event risks in patients with metabolic syndrome at high cardiovascular risk (HCR-MS).
  Participants will adhere to the study protocol, attending regular visits and examinations to assess efficacy and safety.
  Interventions: Drug: Participants will receive Tongmai Jiangtang Capsule (TJC) in addition to standard treatment.
- Control Group (Placebo Group) (Placebo Comparator): Participants in this Arm will receive a placebo capsule that is identical in appearance, size, color, formulation, weight, taste, and smell to TJC, in addition to standard treatment.
  Dosage: Three placebo capsules, three times daily (tid), taken orally. Duration: The intervention period is 26 weeks, followed by a 26-week follow-up. Objective: This Arm serves as a control to compare the efficacy of TJC against a placebo.
  Participants will adhere to the study protocol, attending regular visits and examinations to assess the efficacy and safety of the placebo.
  Interventions: Drug: A placebo capsule that is identical in appearance, size, color, formulation, weight, taste, and smell to TJC

INTERVENTIONS:
Drug: Participants will receive Tongmai Jiangtang Capsule (TJC) in addition to standard treatment. — Intervention Agent: The study employs Tongmai Jiangtang Capsule (TJC), a traditional Chinese medicine compound formulated based on TCM theory. It has the functions of Nourishing Yin, clearing heat and activating blood circulation, and can comprehensively regulate glucose and lipid metabolism as well as improve cardiovascular and cerebrovascular functions.
  Intervention Population: The study focuses on patients with metabolic syndrome at high cardiovascular and cerebrovascular risk (HCR-MS) who meet the TCM criteria for "Qi-deficiency and Blood Stasis syndrome," reflecting personalized and precision intervention.
  Intervention Design: A long-term study design with 26 weeks of intervention followed by 26 weeks of follow-up is adopted to comprehensively assess the short-term efficacy and long-term cardiovascular benefits of TJC.
  Control Design: The study employs a double-blind, randomized, placebo-controlled method.
  Arms: Experimental Group (Tongmai Jiangtang Capsule Group)
Drug: A placebo capsule that is identical in appearance, size, color, formulation, weight, taste, and smell to TJC — Participants in this Arm will receive a placebo capsule that is identical in appearance, size, color, formulation, weight, taste, and smell to TJC, in addition to standard treatment.
  Arms: Control Group (Placebo Group)

SUMMARY:
1. Conduct a large-sample, multicenter, superiority, double-blind, randomized controlled clinical trial to verify the efficacy of TJC in reducing the risk of cardiovascular and cerebrovascular events in patients with metabolic syndrome at high cardiovascular and cerebrovascular risk (HCR-MS).
2. Further construct an evaluation system for the long-term cardiovascular and cerebrovascular benefits of traditional Chinese medicine in regulating glucose and lipid metabolism through the evaluative study of the cardiovascular and cerebrovascular benefits of TJC.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be aged ≥65 years.
* Participants must meet the diagnostic criteria for metabolic syndrome according to the 2020 Chinese Type 2 Diabetes Prevention Guidelines, which includes at least three of the following criteria:①Central obesity: Waist circumference ≥90 cm for men, ≥85 cm for women.②Hyperglycemia: Fasting blood glucose ≥6.1 mmol/L or 2-hour post-load glucose ≥7.8 mmol/L, or a confirmed diagnosis of diabetes with ongoing treatment.③Hypertension: Blood pressure ≥130/85 mmHg or a confirmed diagnosis of hypertension with ongoing treatment.④Elevated triglycerides (TG): ⑤Fasting TG ≥1.70 mmol/L.

Low HDL cholesterol: Fasting HDL-C <1.04 mmol/L.

* Participants must meet the criteria for "Qi-deficiency and Blood Stasis" syndrome, which includes specific symptoms and signs such as fatigue, shortness of breath, stabbing pain, ecchymosis, and a tongue with purple discoloration or petechiae.
* High Cardiovascular Risk: Participants must have at least one of the following:

  * History of myocardial infarction.

    * History of stroke or transient ischemic attack. ③History of coronary, carotid, or peripheral artery revascularization.

      * Coronary, carotid, or lower limb artery stenosis >50%. ⑤Positive exercise stress test or documented symptomatic coronary heart disease, or unstable angina with ECG changes.

        * Chronic heart failure (NYHA Class II-III). ⑦Chronic kidney disease (eGFR <60 ml/min/1.73m²).

Exclusion Criteria:

* Secondary Abnormalities: Secondary abnormalities in lipids, blood pressure, or blood glucose.
* Type 1 Diabetes: Participants with Type 1 diabetes mellitus.
* Special Populations: Pregnant or breastfeeding individuals, or those with a history of allergy to the study medication.
* Recent Acute Events: Acute coronary or cerebrovascular events within the past 14 days.
* Upcoming Revascularization: Planned coronary, carotid, or peripheral artery revascularization.
* Severe Heart Failure: Chronic heart failure (NYHA Class IV).
* End-Stage Liver Disease: Participants with end-stage liver disease.
* Solid Organ Transplantation: History of solid organ transplantation or awaiting solid organ transplantation.
* Malignant Tumors: Participants with a history of malignant tumors.
* Other Serious Conditions: Any other serious medical conditions that may interfere with the study or pose a risk to the participant.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | From enrollment to the next 52 weeks
  sudden cardiac death or death due to myocardial infarction, heart failure, stroke, or other cardiovascular causes.
Non-fatal myocardial infarction | From enrollment to the next 52 weeks
  Including spontaneous, STEMI, NSTEMI, PCI-related, CABG-related, and silent acute myocardial infarction
Non-fatal stroke | From enrollment to the next 52 weeks
  Meet any one of the following criteria:
  * Acute neurological dysfunction documented by CT/MRI, attributable to vascular causes with other etiologies excluded; ② Transient ischemic attack (TIA) lasting <24 hours; ③ Microhemorrhage: Round hypointense lesions <5-10 mm on MRI.

SECONDARY OUTCOMES:
Composite cardiovascular outcomes | From enrollment to the next 52 weeks
  death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, coronary revascularization, or hospitalization for unstable angina or heart failure
All-cause mortality | From enrollment to the next 52 weeks
  Any cause of death
Renal and diabetes-related microvascular composite outcomes | From enrollment to the next 52 weeks
  Including renal outcomes or diabetic retinopathy outcomes
blood glucose | From enrollment to the next 52 weeks
  Including fasting plasma glucose (FPG), 2-hour postprandial blood glucose (2h PPG), and glycated hemoglobin (HbA1c).
lipids | From enrollment to the next 52 weeks
  Including total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C).
Blood pressure | From enrollment to the next 52 weeks
  Including systolic blood pressure and systolic blood pressure
BMI | From enrollment to the next 52 weeks
  Body Mass Index
waist-to-hip ratio | From enrollment to the next 52 weeks
  waist-to-hip ratio
HOMA-IR | From enrollment to the next 52 weeks
  HOMA-IR=(Fasting Glucose (mmol/L)×Fasting Insulin (μU/mL))/22.5
Body fat analysis | From enrollment to the next 52 weeks
  Including Body Fat Percentage (BFP) and Visceral Fat Index (VFI)
Vitamin D levels | From enrollment to the next 52 weeks
  Vitamin D levels
Assessment of peripheral vascular status | From enrollment to the next 52 weeks
  Assessment of plaque or stenosis in the common carotid artery
Cardiac function | From enrollment to the next 52 weeks
  Including Cardiac Enzymes, Troponin, BNP, Ejection Fraction (EF), Left Ventricular Myocardial Thickness, and Interventricular Septal Thickness.
Cardiovascular risk indices | From enrollment to the next 52 weeks
  Including the China-PAR Score, Framingham Risk Score, and QRISK3 Score.
Traditional Chinese medicine symptom scores | From enrollment to the next 52 weeks
  Including symptoms related to observation, hearing, questioning, and palpation.
Quality of life scores. | From enrollment to the next 52 weeks
  The Short-From-36 Health Survey, SF-36
Omics analysis | From enrollment to the next 52 weeks
  Including transcriptomics, proteomics, untargeted metabolomics, and microbiome analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Marso SP, Poulter NR, Nissen SE, Nauck MA, Zinman B, Daniels GH, Pocock S, Steinberg WM, Bergenstal RM, Mann JF, Ravn LS, Frandsen KB, Moses AC, Buse JB. Design of the liraglutide effect and action in diabetes: evaluation of cardiovascular outcome results (LEADER) trial. Am Heart J. 2013 Nov;166(5):823-30.e5. doi: 10.1016/j.ahj.2013.07.012. Epub 2013 Oct 2. PMID 24176437